CLINICAL TRIAL: NCT06651216
Title: Impact of Breast Milk miRNAs on the Infant Gut Microbiota
Acronym: MiMilk
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP240711; IDRCB: 2024-A01059-38 (Registry Identifier: ANSM)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Breast Milk; Stools
MeSH Terms: interventions — Occult Blood

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool and breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast feeding: Exclusively breastfed infants for 2 months
  Interventions: Other: Stool analysis; Other: breast milk analysis
- Non breast feeding: Infants exclusively fed with formula milk
  Interventions: Other: Stool analysis

INTERVENTIONS:
Other: Stool analysis — Analysis of infant fecal microbiota
Other: breast milk analysis — Analysis of the effect of breast milk miRNAs on infant fecal microbiota
  Groups: Breast feeding

SUMMARY:
The first 1000 days of life are a critical period for future health. A healthy gut microbiota (GM) is essential for preventing both short-term and long-term health issues. Breast milk (BM) plays a key role in establishing the GM, as, unlike formula milk, it contains miRNAs that may interact with and modulate the microbiota.

Primary Objective: To study the effect of BM on the composition of fecal miRNAs in exclusively breastfed infants compared to those fed with formula milk at different times (D10, D30, D60, M6, M12).

Secondary Objectives:

Analyze the effect of BM miRNAs on infant fecal microbiota, taking environmental confounding factors into account.

Study the influence of BM microbiota on miRNA profiles in the milk. Examine the effect of BM microbiota on the infants' gut microbiota. Explore the links between BM miRNAs, infant gut microbiota, and intestinal inflammation.

DETAILED DESCRIPTION:
The first 1,000 days of life are a critical period that significantly contributes to the programming of an individual's health. It is increasingly evident that establishing a healthy gut microbiota (GM) plays an important role in preventing both short- and long-term health issues.

Among the factors influencing the establishment of the infant's gut microbiota, breast milk (BM) plays a fundamental role. Unlike formula milk, breast milk contains miRNAs that are potential mediators of the interactions between the host and the microbiota. Thus, we hypothesize that miRNAs from breast milk may be present in the infant's luminal content and interact with their microbiota, thereby modulating it.

Main Objective: Explore the effect of breast milk on the composition of fecal miRNAs in infants.

Primary Evaluation Criterion: Profiles and quantities of miRNAs at different time points (D10, D30, D60, M6, and M12) in the stools of exclusively breastfed infants compared to those fed with formula milk.

Secondary Objectives:

Study the effect of miRNAs from breast milk on the composition of the infant's fecal microbiota, considering environmental confounding factors, including the composition of maternal microbiota.

Investigate the effect of breast milk microbiota on the miRNA profiles present in the milk.

Study the effect of breast milk microbiota on the gut microbiota of infants. Explore the links between breast milk miRNAs, the infant's gut microbiota, and intestinal inflammation in infants.

Secondary Evaluation Criteria:

Correlations between breast milk miRNA profiles from D1 to D60 and the gut microbiota of breastfed infants from D1 to M12.

Correlations between the breast milk microbiota and the breast milk miRNA profiles from D1 to D60.

Correlations between breast milk microbiota from D1 to D60 and the infant fecal microbiota from D1 to M12.

Direct correlations between (1) breast milk miRNAs and the measurement of fecal calprotectin in infants from D1 to D60, and (2) the infant's gut microbiota and fecal calprotectin in infants from D1 to D60.

To address the research question, we plan to include 200 mother-infant dyads. Our goal is to have 30 dyads with exclusive breastfeeding for at least two months, and 30 dyads where the infant will not have received any breast milk. Each dyad will participate in the study for a period of 12 months, and the recruitment phase will last for 18 months.

At the infant's birth, we will collect stool samples from both the mother and the infant, as well as a breast milk sample from the mother.

At 10, 30, and 60 days after the infant's birth, we will request both a breast milk sample from the mother and a stool sample from the infant.

At 6 and 12 months, only a stool sample from the infant will be collected. During each visit, a clinical research coordinator will contact the mothers to gather information about both their health and diet, as well as their infant's health and diet.

Analysis of miRNAs in Breast Milk and Stool Samples: miRNAs will be extracted from infant stool samples and breast milk using next-generation Illumina sequencing (NGS). The top 10 most abundant miRNAs will then be validated through qPCR. The overall miRNA profiles will be analyzed using Principal Coordinate Analysis (PCoA).

Analysis of Gut and Breast Milk Microbiota: Stool and breast milk samples will be used for 16S rRNA gene sequencing to analyze the microbial composition. Microbiota profiles will also be examined using Principal Coordinate Analysis (PCoA).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the 3rd trimester of pregnancy (3T) with a normal course of pregnancy up to 39 weeks consulting for the monitoring visit at the Robert-Debré hospital.
* Patients who did not receive antibiotic treatment or probiotics in 3T.
* Patient with a negative PV for Strepto B
* Patients who do not have complications such as pre-eclampsia or gestational diabetes.
* Breastfeeding (+/- milk pump) or exclusive artificial breastfeeding.
* No opposition from the mother
* Ability to master the French language required.
* Freezer at home.
* Affiliation to a social security scheme.

Exclusion Criteria:

* Cesarean delivery
* Perinatal pathologies (Anoxia, IUGR, etc.)
* Neonatal pathologies (FGR, malformations, etc.)
* Initial choice of mixed breastfeeding
* Patient under AME (State Medical Aid)Critères d'exclusions :
* Antibiotics for the mother or child before day 60
* Antifungal for the mother or child before day 60
* Complete cessation of breastfeeding before day 60

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Mother-child dyad in good health from birth
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Explore the effect of breast milk on the composition of fecal miRNAs in infants | 12 months
  profiles and quantities of miRNAs at different times (D10, D30, D60, M6, and M12) in the stools of exclusively breastfed infants compared to those fed with formula milk

CONTACTS AND LOCATIONS:
Overall Officials: Alexis MOSCA, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital Assistance Publique Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided